CLINICAL TRIAL: NCT00340912
Title: Use of Biopsy Punch for Skin Biopsies for Fibroblasts Culturing
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999880215; OH88-DK-0215
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-01

CONDITIONS: Fibroblasts
Keywords: Skin Biopsy

SUMMARY:
Fibroblasts can be cultured from human skin biopsies using fetal bovine serum and artificial growth medium. Fibroblasts cultured in this way retain the genetic characteristics of their donor but can be used for experiments where study conditions are much more precisely controlled than they can be in in vivo studies. We plan to culture fibroblasts from Pima Indians for two purposes. Firstly, to look for an in vitro system to measure insulin resistance, the underlying abnormality in Pima diabetics. Secondly, to look for biochemical markers of diabetes or obesity in Pimas employing two dimensional electrophoresis techniques.

DETAILED DESCRIPTION:
Fibroblasts can be cultured from human skin biopsies using fetal bovine serum and artificial growth medium. Fibroblasts cultured in this way retain the genetic characteristics of their donor but can be used for experiments where study conditions are much more precisely controlled than they can be in in vivo studies. We plan to culture fibroblasts from Pima Indians for two purposes: 1) to look for an in vitro system to measure insulin resistance, the underlying abnormality in Pima diabetics; and 2) to look for biochemical markers of diabetes or obesity in Pimas employing two-dimensional electrophoresis techniques.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include Pima Indians who do not meet any of the exclusion criteria.

EXCLUSION CRITERIA:

We will exclude any seriously ill individuals, any known to have a bleeding diathesis or to be immunosuppressed or subjects who are carriers of HIV or HBV.

Children will be excluded, as the age range for this study's participants is 18-50.

Pregnant women will be excluded on the basis of a urinary pregnancy test.

All other subjects are potentially included.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500
Dates: Start 1988-12-07; Primary Completion 1988-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States